CLINICAL TRIAL: NCT03065465
Title: Randomized Controlled Trial (RCT) of Standard Endoscopic Hemostasis Compared to OVESCO for Severe Non-variceal UGI Hemorrhage
Brief Title: Standard Endoscopic Hemostasis Versus OVESCO Severe Non-variceal UGI Hemorrhage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CURE Digestive Diseases Research Center (Other)
Collaborators: University of California, Los Angeles (Other); VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OVESCO
Record Dates: First submitted 2016-11-29; First posted 2017-02-28 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-01

CONDITIONS: Upper Gastrointestinal Hemorrhage
Keywords: Upper GI hemorrhage; Stigmata of recent hemorrhage; Ulcers; Dieulafoy's lesions
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard endoscopic treatment (Other): For those assigned to the standard endoscopy group, endoscopic hemostasis is performed using usual CURE hemostasis therapy for the focal GI lesions: injection of dilute (e.g. 1: 20,000) epinephrine (in 1-2 cc aliquots in 4 quadrants next to the SRH) of active bleeding or adherent clots (prior to snaring them off); coaptive coagulation with multipolar electrocautery (MPEC) probe and/or standard through the endoscope hemoclips along the course of the underlying artery as detected by DEP. Hemostasis is performed until active bleeding stops and/or the SRH is obliterated. Residual blood flow after visually guided hemostasis is recorded, but not used as a guide for additional hemostasis in this study.
  Interventions: Other: Standard endoscopic treatment
- Over-the-scope hemoclipping device (Experimental): For those assigned OTSC, prior to use of the OTSC in UGI lesions with active bleeding or adherent clots, dilute epinephrine (1: 20,000) is injected around the SRH in 1-2 cc aliquots and the clots are cold guillotined off, as previously described (2, 4, 17). As a brief additional description, after initial diagnosis and preparation of the lesion and SRH (as described for standard hemostasis), the therapeutic sized endoscope is removed and this or a diagnostic panendoscope will be affixed with the OTSC of appropriate size for the endoscope and the target lesion. The endoscope is re-introduced and passed to the bleeding site. The SRH is centered in the field of view and within the cap of the OTSC device. Using high suctioning and firm pressure to center the SRH, the lesion and SRH is captured into the cap and the OTSC is deployed by rotating the handle and thereby compressing the bleeding lesion and surrounding tissue with mechanical hemostasis.
  Interventions: Device: Over-the-scope hemoclipping device

INTERVENTIONS:
Device: Over-the-scope hemoclipping device — A endoscopic entrapment of tissue for control of bleeding or other applications.
  Other Names: OTSC clip
  Arms: Over-the-scope hemoclipping device
Other: Standard endoscopic treatment — Standard therapy includes injection of dilute epinephrine, thermal coagulation with multipolar electrocautery (MPEC) probe, and/or hemoclips.
  Arms: Standard endoscopic treatment

SUMMARY:
The primary specific aim is to perform a randomized controlled trial (RCT) to compare 30 day rebleed rates and other clinical outcomes of patients with severe, non-variceal upper GI hemorrhage (NVUGIH) - ulcers and Dieulafoy's lesions who are randomized as initial treatment with the new large over-the-scope-clip device for endoscopic hemostasis versus standard endoscopic hemostasis.

DETAILED DESCRIPTION:
Upper GI Hemorrhage (UGIH) causes significant morbidity and mortality, although endoscopic hemostasis has revolutionized management of these patients. Despite standard endoscopic treatment and high dose proton pump infusions, 25% - 30% of high risk patients with UGIB from ulcers or other non-variceal UGI lesions (NVUGI) had recurrent bleeding in a recent RCT and cohort studies by our group. Potential risk factors for NVUGI rebleeding were large ulcers (≥ 15 mm), fibrotic bases, Dieulafoy's lesions, anastomotic ulcers, coagulopathies, cirrhosis, other severe co-morbidities and residual arterial blood flow under stigmata of recent hemorrhage (SRH) after endoscopic treatment. Such patients with rebleeding after standard endoscopic hemostasis usually required angiography (by interventional radiologists-IR) or surgery for definitive hemostasis. A new, large, FDA approved, over-the-scope hemoclipping device (OTSC® System OVESCO Endoscopy, Tübingen, Germany) can capture larger amounts of tissue and underlying arteries than standard hemoclips and potentially can improve endoscopic hemostasis of such bleeding lesions.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from the patient or a surrogate.
* Clinical evidence of severe UGIB.
* Presence of a benign appearing peptic ulcer, anastomotic ulcer, or Dieulafoy's lesion, with some SRH on endoscopy.
* Severe upper GI bleeding.
* Life expectancy of at least 30 days based on lack of severe or terminal comorbidity as judged by the generalist or subspecialist caring for the patient.

Exclusion Criteria:

* Patients who are do-not-resuscitate (DNR) that is not reversible, uncooperative, refuse to participate, or are unable to give consent personally or through a legal surrogate.
* Active GI malignancy, under treatment but not in remission.
* Acute hypovolemic shock that is unresponsive to transfusion of 5 or more units of red blood cells (RBC's) or requires continuous intravenous vasopressor infusion for blood pressure support.
* ASA (American Society of Anesthesiology) class V or higher, moribund, or with a very poor prognosis and expected survival <30 days.
* Severe coagulopathy or thrombocytopenia despite attempted reversal with transfusion of blood products (e.g persistent International Normalized Ratio [INR] >2.0, platelet count <20,000, a Partial Thromboplastin Time [PTT] greater than 2x upper limit of normal).
* Absolute contraindication to urgent endoscopy (such as suspected perforated viscus, or peritonitis).
* Stricture of the esophagus or pylorus that can not be dilated or precludes passage of a diagnostic sized endoscope and/or the GI endoscope with an 11, 3a OTSC device attached.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2015-11-15; Primary Completion 2024-12-24 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
The rebleeding rate of non-variceal focal UGI lesions | Outcome measure will be assessed at 30 days after participants are enrolled
  The investigators will compare the rebleeding rate at 30 days follow up in the two treatment groups for all patients, ulcer patients only, and also patients with major stigmata of hemorrhage vs. lesser stigmata (oozing or flat spots).

SECONDARY OUTCOMES:
Obliteration rates of underlying arterial blood flow (detected by Doppler endoscopic probe) | Outcome measure will be assessed at 30 days after the endoscopy treatment is completed
  The investigators will use the Doppler endoscopic probe to measure the blood flow before and after the application of over-the-hemoclipping device and standard endoscopic hemostasis.
Rates of surgery or IR, complications, and death | Outcome measure will be assessed at 30 days after participants are enrolled
  The investigators will compare the rates of surgery or IR, complications, transfusion, hospital stays, and death at 30 days for the two treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis M Jensen, MD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laine L, Jensen DM. Management of patients with ulcer bleeding. Am J Gastroenterol. 2012 Mar;107(3):345-60; quiz 361. doi: 10.1038/ajg.2011.480. Epub 2012 Feb 7. PMID 22310222
- [Background] Camus M, Jensen DM, Kovacs TO, Jensen ME, Markovic D, Gornbein J. Independent risk factors of 30-day outcomes in 1264 patients with peptic ulcer bleeding in the USA: large ulcers do worse. Aliment Pharmacol Ther. 2016 May;43(10):1080-9. doi: 10.1111/apt.13591. Epub 2016 Mar 22. PMID 27000531
- [Background] Jensen DM, Kovacs TOG, Ohning GV, Ghassemi K, Machicado GA, Dulai GS, Sedarat A, Jutabha R, Gornbein J. Doppler Endoscopic Probe Monitoring of Blood Flow Improves Risk Stratification and Outcomes of Patients With Severe Nonvariceal Upper Gastrointestinal Hemorrhage. Gastroenterology. 2017 May;152(6):1310-1318.e1. doi: 10.1053/j.gastro.2017.01.042. Epub 2017 Feb 4. PMID 28167214
- [Background] Schmidt A, Golder S, Goetz M, Meining A, Lau J, von Delius S, Escher M, Hoffmann A, Wiest R, Messmann H, Kratt T, Walter B, Bettinger D, Caca K. Over-the-Scope Clips Are More Effective Than Standard Endoscopic Therapy for Patients With Recurrent Bleeding of Peptic Ulcers. Gastroenterology. 2018 Sep;155(3):674-686.e6. doi: 10.1053/j.gastro.2018.05.037. Epub 2018 May 24. PMID 29803838
- [Background] Nishiyama N, Mori H, Kobara H, Rafiq K, Fujihara S, Kobayashi M, Oryu M, Masaki T. Efficacy and safety of over-the-scope clip: including complications after endoscopic submucosal dissection. World J Gastroenterol. 2013 May 14;19(18):2752-60. doi: 10.3748/wjg.v19.i18.2752. PMID 23687412
- [Background] Monkemuller K, Peter S, Toshniwal J, Popa D, Zabielski M, Stahl RD, Ramesh J, Wilcox CM. Multipurpose use of the 'bear claw' (over-the-scope-clip system) to treat endoluminal gastrointestinal disorders. Dig Endosc. 2014 May;26(3):350-7. doi: 10.1111/den.12145. Epub 2013 Jul 16. PMID 23855514
- [Background] Kirschniak A, Kratt T, Stuker D, Braun A, Schurr MO, Konigsrainer A. A new endoscopic over-the-scope clip system for treatment of lesions and bleeding in the GI tract: first clinical experiences. Gastrointest Endosc. 2007 Jul;66(1):162-7. doi: 10.1016/j.gie.2007.01.034. PMID 17591492
- [Background] Manta R, Galloro G, Mangiavillano B, Conigliaro R, Pasquale L, Arezzo A, Masci E, Bassotti G, Frazzoni M. Over-the-scope clip (OTSC) represents an effective endoscopic treatment for acute GI bleeding after failure of conventional techniques. Surg Endosc. 2013 Sep;27(9):3162-4. doi: 10.1007/s00464-013-2871-1. Epub 2013 Feb 23. PMID 23436101
- [Background] Richter-Schrag HJ, Glatz T, Walker C, Fischer A, Thimme R. First-line endoscopic treatment with over-the-scope clips significantly improves the primary failure and rebleeding rates in high-risk gastrointestinal bleeding: A single-center experience with 100 cases. World J Gastroenterol. 2016 Nov 7;22(41):9162-9171. doi: 10.3748/wjg.v22.i41.9162. PMID 27895403
- [Background] Wedi E, von Renteln D, Gonzalez S, Tkachenko O, Jung C, Orkut S, Roth V, Tumay S, Hochberger J. Use of the over-the-scope-clip (OTSC) in non-variceal upper gastrointestinal bleeding in patients with severe cardiovascular comorbidities: a retrospective study. Endosc Int Open. 2017 Sep;5(9):E875-E882. doi: 10.1055/s-0043-105496. Epub 2017 Sep 12. PMID 28924593
- [Background] Golder S, Neuhas L, Freuer D, Probst A, Ebigbo A, Braun G, Brueckner J, Stueckle J, Meier A, Messmann H. Over-the-scope clip in peptic ulcer bleeding: clinical success in primary and secondary treatment and factors associated with treatment failure. Endosc Int Open. 2019 Jun;7(6):E846-E854. doi: 10.1055/a-0898-3357. Epub 2019 Jun 13. PMID 31206010
- [Background] Wedi E, Fischer A, Hochberger J, Jung C, Orkut S, Richter-Schrag HJ. Multicenter evaluation of first-line endoscopic treatment with the OTSC in acute non-variceal upper gastrointestinal bleeding and comparison with the Rockall cohort: the FLETRock study. Surg Endosc. 2018 Jan;32(1):307-314. doi: 10.1007/s00464-017-5678-7. Epub 2017 Jun 27. PMID 28656336
- [Background] Brandler J, Baruah A, Zeb M, Mehfooz A, Pophali P, Wong Kee Song L, AbuDayyeh B, Gostout C, Mara K, Dierkhising R, Buttar N. Efficacy of Over-the-Scope Clips in Management of High-Risk Gastrointestinal Bleeding. Clin Gastroenterol Hepatol. 2018 May;16(5):690-696.e1. doi: 10.1016/j.cgh.2017.07.020. Epub 2017 Jul 26. PMID 28756055
- [Background] Chandrasekar VT, Desai M, Aziz M, Patel HK, Gorrepati VS, Jegadeesan R, Rai T, Sathyamurthy A, Murino A, Hassan C, Repici A, Sharma P. Efficacy and safety of over-the-scope clips for gastrointestinal bleeding: a systematic review and meta-analysis. Endoscopy. 2019 Oct;51(10):941-949. doi: 10.1055/a-0994-4361. Epub 2019 Aug 30. PMID 31470449
- [Background] Jensen DM, Ohning GV, Kovacs TO, Ghassemi KA, Jutabha R, Dulai GS, Machicado GA. Doppler endoscopic probe as a guide to risk stratification and definitive hemostasis of peptic ulcer bleeding. Gastrointest Endosc. 2016 Jan;83(1):129-36. doi: 10.1016/j.gie.2015.07.012. Epub 2015 Aug 28. PMID 26318834
- [Background] Jensen DM, Kovacs TO, Jutabha R, Machicado GA, Gralnek IM, Savides TJ, Smith J, Jensen ME, Alofaituli G, Gornbein J. Randomized trial of medical or endoscopic therapy to prevent recurrent ulcer hemorrhage in patients with adherent clots. Gastroenterology. 2002 Aug;123(2):407-13. doi: 10.1053/gast.2002.34782. PMID 12145792
- [Derived] Jensen DM, Kovacs T, Ghassemi KA, Kaneshiro M, Gornbein J. Randomized Controlled Trial of Over-the-Scope Clip as Initial Treatment of Severe Nonvariceal Upper Gastrointestinal Bleeding. Clin Gastroenterol Hepatol. 2021 Nov;19(11):2315-2323.e2. doi: 10.1016/j.cgh.2020.08.046. Epub 2020 Aug 20. PMID 32828873